CLINICAL TRIAL: NCT06096051
Title: Evaluation of 4-Factor PCC in DOAC-associated Intracranial Hemorrhage
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 027.PHA.2023.A
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-08

CONDITIONS: Intracranial Hemorrhage
MeSH Terms: conditions — Intracranial Hemorrhages

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Use of fixed-dosed 4F-PCC — Determine if fixed-dose 4F-PCC is safe and effective in patients with DOAC-associated ICH when compared to weight-based dosing.

SUMMARY:
Intracranial hemorrhage (ICH) can occur due to traumatic and spontaneous events.1 The incidence of non-traumatic, spontaneous ICH is approximately 40,000 to 67,000 cases per year while the incidence of traumatic brain injury (TBI) is nearly 1.7 million annually

DETAILED DESCRIPTION:
The authors found that AC use preinjury was associated with ICH progression, immediate neurosurgery intervention, and death after initial scan. AC use has also been associated with worse functional outcomes, and patients are less likely to be discharged home compared to those without AC use prior to injury.6 With increasing prevalence of AC, hospitals are seeing admissions for ICH, making knowledge of optimal AC reversal essential.

ELIGIBILITY:
Inclusion Criteria:

* • ≥18 years of age

  * ICH (traumatic and spontaneous)
  * Administration of at least one dose of 4F-PCC
  * Admitted to the MHS between July 1, 2018 and May 30, 2023
  * Rivaroxaban or apixaban use prior to admission

Exclusion Criteria:

* • Warfarin or dabigatran use prior to admission

  * Prisoners
  * Pregnancy
  * <18 years of age

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients 18 years of age
  * ICH (traumatic and spontaneous)
  * Administration of at least one dose of 4F-PCC
  * Admitted to the MHS between July 1, 2018 and May 30, 2023
  * Rivaroxaban or apixaban use prior to admission
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2024-07-13 (Estimated); Study Completion 2024-07-13 (Estimated)

PRIMARY OUTCOMES:
Determine safety and effectiveness of 4F-PCC | 12 hours
  fixed-dose 4F-PCC is safe and effective in patients with DOAC-associated ICH when compared to weight-based dosing.

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Reiter, PharmD, Principal Investigator — Methodist Midlothian Medical Center
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Study data or any protected health information will not be shared with anyone that is not delegated to the study. The PI is committed to disseminate research results in a timely fashion. Sharing of results generated by the data analysis during the course of the project will be through presentation at national scientific meetings and/or publication in open access journals. All information obtained will be source de-identified and presented on a large scale and not traceable to any one particular individual
Time Frame: 2 years

REFERENCES:
- [Background] Tenny S, Das JM, Thorell W. Intracranial Hemorrhage. 2024 Feb 17. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK470242/ PMID 29262016